CLINICAL TRIAL: NCT01397513
Title: Effects of Low and High Doses of Aspirin Treatment on Fibrin Network Formation in Patients With Type 1 Diabetes and Possible Influence of the Glycemic Control.
Brief Title: Effects of Aspirin Treatment on Fibrin Network Formation in Patients With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Gun Jörneskog, Karolinska Institutet, Department of Clinical Sciences, Danderyd Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 151:2005/76316; 2005/1403-31/2 (Other: Ethics Committe in Stockholm)
Record Dates: First submitted 2011-07-14; First posted 2011-07-19 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2006-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Fibrin network structure; Aspirin treatment; Platelet microparticles
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin 75mg (Active Comparator)
  Interventions: Drug: Aspirin
- Aspirin 320mg (Active Comparator)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Tablets, 75 or 320mg once daily for 4 weeks. A 4-week wash-out period separated the two treatment periods.
  Other Names: Trombyl

SUMMARY:
The fibrin network is an important component of an arterial thrombus and its structure influences the degradation of the formed clot. A tighter and less permeable fibrin network, which is less susceptible to fibrinolysis, is formed in patients with manifest cardiovascular disease (CVD) or conditions associated with increased risk of atherothrombotic complications. In a previous study we have shown reduced fibrin network permeability in patients with type 1 diabetes, which may contribute to their increased risk of CVD. Low dose aspirin treatment is standard in management of CVD; however, the effect seems reduced in patients with diabetes. Our previous studies have shown that aspirin treatment alters the fibrin network in non-diabetic individuals and increases the fibrin network permeability. The effect of aspirin on fibrin network formation in patients with diabetes is unclear.

We hypothesized that patients with type 1 diabetes might need higher doses of aspirin than the recommended low dose (75mg) treatment to gain effects on fibrin network permeability, and that the effects of aspirin treatment on fibrin network in these patients are influenced by the glycemic control.

DETAILED DESCRIPTION:
Diabetes is associated with increased platelet activation, elevated plasma fibrinogen levels and impaired fibrinolysis, factors which may contribute to the elevated risk of cardiovascular disease (CVD) in these patients. Increased platelet activation in patients with diabetes is reflected by elevated levels of platelet microparticles, which are small circulating procoagulant vesicles shed from the platelet membrane upon activation. CVD in these patients may start as early as in the age of 25-30 years and the course is often aggressive and with poor prognosis. Treatment with a daily low dose of acetylsalicylic acid (aspirin 75 mg) is one of the cornerstones in management of CVD in non-diabetic patients; however, the effect seems reduced in patients with diabetes. The mechanisms behind this treatment failure with aspirin in diabetes patients are unclear. Aspirin is a complex drug with multiple effects. The most well known is acetylation and inhibition of platelet cyclooxygenase (COX), but COX-independent mechanisms may also of importance in protection of cardiovascular complications. One such mechanism is alteration of the fibrin/fibrinogen properties and the fibrin network structure, possibly through acetylation of the lysine residues in the fibrinogen molecule involved in crosslinking of fibrin. The fibrin network structure seems important in development of atherothrombotic events, as individuals at high risk of CVD, including patients with type 1 diabetes, as well as patients with manifest CVD have a tighter and less permeable fibrin network structure. The altered fibrin network in patients with type 1 diabetes may in part be due to increased fibrinogen glycation, which may occur on lysine residues. Treatment with aspirin increases fibrin network permeability in non-diabetic subjects. However, the effect of aspirin on fibrin network permeability in patients with diabetes is unclear. Possible competition between acetylation and glycation on lysine residues in the fibrinogen molecule might contribute to the reduced preventive effect of aspirin in management of CVD in patients with diabetes and higher doses of aspirin might therefore be required in these patients.

Our hypothesis was that glycation and acetylation occur at the same binding sites in the fibrinogen molecule. Thus, poor glycemic control and increased glycation may lead to lower acetylation of the fibrinogen molecule than during good glycemic control in turn leading to an altered fibrin network.

The aims of the present study were to analyse the effects of low (75 mg) and high dose (320 mg) aspirin treatment on fibrin network formation in patients with type 1 diabetes (primary aim), and to investigate the possible influence of the glycemic control (secondary aim). As platelet microparticles may influence the fibrin formation [17, 18] and since aspirin has well-known effects on platelet function, we also measured plasma concentrations of platelet microparticles.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, type 1
* Levels of HbA1C (glycated hemoglobin) <7.4% (NGSP standard)
* Levels of HbA1C >8.4% (NGSP standard)

Exclusion Criteria:

* Prior aspirin treatment
* Treatment with anticoagulant drugs
* Ongoing treatment with NSAIDs or other antiplatelet drugs
* A history of macrovascular disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-03; Primary Completion 2010-07 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Fibrin network permeability | At the start and end of each 4-week treatment period
  Changes in fibrin network permeability after 4 weeks of treatment with either aspirin 75 or 320mg.

SECONDARY OUTCOMES:
Fibrin network permeability | At the start and end of each 4-week treatment period
  Subgroup analyses comparing the treatment effects of aspirin 75 or 320mg on fibrin network permeability in patients with good and poor glycemic control, respectively.
Platelet microparticles | At the start and end of each 4-week treatment period
  Changes in plasma concentrations of platelet microparticles after 4 weeks of treatment with either aspirin 75 or 320mg.

CONTACTS AND LOCATIONS:
Overall Officials: Gun Jörneskog, MD PhD, Principal Investigator — Karolinska Institutet, Department of Clinical Sciences, Danderyd Hospital
Locations (1):
- Karolinska Institutet, Department of Clinical Sciences, Danderyd Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Collet JP, Park D, Lesty C, Soria J, Soria C, Montalescot G, Weisel JW. Influence of fibrin network conformation and fibrin fiber diameter on fibrinolysis speed: dynamic and structural approaches by confocal microscopy. Arterioscler Thromb Vasc Biol. 2000 May;20(5):1354-61. doi: 10.1161/01.atv.20.5.1354. PMID 10807754
- [Background] Collet JP, Allali Y, Lesty C, Tanguy ML, Silvain J, Ankri A, Blanchet B, Dumaine R, Gianetti J, Payot L, Weisel JW, Montalescot G. Altered fibrin architecture is associated with hypofibrinolysis and premature coronary atherothrombosis. Arterioscler Thromb Vasc Biol. 2006 Nov;26(11):2567-73. doi: 10.1161/01.ATV.0000241589.52950.4c. Epub 2006 Aug 17. PMID 16917107
- [Background] Rooth E, Wallen NH, Blomback M, He S. Decreased fibrin network permeability and impaired fibrinolysis in the acute and convalescent phase of ischemic stroke. Thromb Res. 2011 Jan;127(1):51-6. doi: 10.1016/j.thromres.2010.09.011. Epub 2010 Oct 14. PMID 20950841
- [Background] Colle JP, Mishal Z, Lesty C, Mirshahi M, Peyne J, Baumelou A, Bensman A, Soria J, Soria C. Abnormal fibrin clot architecture in nephrotic patients is related to hypofibrinolysis: influence of plasma biochemical modifications: a possible mechanism for the high thrombotic tendency? Thromb Haemost. 1999 Nov;82(5):1482-9. PMID 10595642
- [Background] Jorneskog G, Egberg N, Fagrell B, Fatah K, Hessel B, Johnsson H, Brismar K, Blomback M. Altered properties of the fibrin gel structure in patients with IDDM. Diabetologia. 1996 Dec;39(12):1519-23. doi: 10.1007/s001250050607. PMID 8960835
- [Background] Cubbon RM, Gale CP, Rajwani A, Abbas A, Morrell C, Das R, Barth JH, Grant PJ, Kearney MT, Hall AS. Aspirin and mortality in patients with diabetes sustaining acute coronary syndrome. Diabetes Care. 2008 Feb;31(2):363-5. doi: 10.2337/dc07-1745. Epub 2007 Oct 24. PMID 17959865
- [Background] Antovic A, Perneby C, Ekman GJ, Wallen HN, Hjemdahl P, Blomback M, He S. Marked increase of fibrin gel permeability with very low dose ASA treatment. Thromb Res. 2005;116(6):509-17. doi: 10.1016/j.thromres.2005.02.007. PMID 16181986
- [Background] Williams S, Fatah K, Hjemdahl P, Blomback M. Better increase in fibrin gel porosity by low dose than intermediate dose acetylsalicylic acid. Eur Heart J. 1998 Nov;19(11):1666-72. doi: 10.1053/euhj.1998.1088. PMID 9857919
- [Background] Yngen M, Ostenson CG, Hu H, Li N, Hjemdahl P, Wallen NH. Enhanced P-selectin expression and increased soluble CD40 Ligand in patients with Type 1 diabetes mellitus and microangiopathy: evidence for platelet hyperactivity and chronic inflammation. Diabetologia. 2004 Mar;47(3):537-540. doi: 10.1007/s00125-004-1352-4. Epub 2004 Feb 13. PMID 14963650
- [Background] Ganda OP, Arkin CF. Hyperfibrinogenemia. An important risk factor for vascular complications in diabetes. Diabetes Care. 1992 Oct;15(10):1245-50. doi: 10.2337/diacare.15.10.1245. PMID 1425083
- [Background] Dunn EJ, Philippou H, Ariens RA, Grant PJ. Molecular mechanisms involved in the resistance of fibrin to clot lysis by plasmin in subjects with type 2 diabetes mellitus. Diabetologia. 2006 May;49(5):1071-80. doi: 10.1007/s00125-006-0197-4. Epub 2006 Mar 16. PMID 16538489
- [Background] Nomura S, Suzuki M, Katsura K, Xie GL, Miyazaki Y, Miyake T, Kido H, Kagawa H, Fukuhara S. Platelet-derived microparticles may influence the development of atherosclerosis in diabetes mellitus. Atherosclerosis. 1995 Aug;116(2):235-40. doi: 10.1016/0021-9150(95)05551-7. PMID 7575778
- [Background] Undas A, Brummel-Ziedins KE, Mann KG. Antithrombotic properties of aspirin and resistance to aspirin: beyond strictly antiplatelet actions. Blood. 2007 Mar 15;109(6):2285-92. doi: 10.1182/blood-2006-01-010645. Epub 2006 Dec 5. PMID 17148593
- [Background] Bjornsson TD, Schneider DE, Berger H Jr. Aspirin acetylates fibrinogen and enhances fibrinolysis. Fibrinolytic effect is independent of changes in plasminogen activator levels. J Pharmacol Exp Ther. 1989 Jul;250(1):154-61. PMID 2746495
- [Background] Lutjens A, te Velde AA, vd Veen EA, vd Meer J. Glycosylation of human fibrinogen in vivo. Diabetologia. 1985 Feb;28(2):87-9. doi: 10.1007/BF00279921. PMID 3920098
- [Background] Ardawi MS, Nasrat HN, Mira SA, Fatani HH. Comparison of glycosylated fibrinogen, albumin, and haemoglobin as indices of blood glucose control in diabetic patients. Diabet Med. 1990 Nov;7(9):819-24. doi: 10.1111/j.1464-5491.1990.tb01499.x. PMID 2148136
- [Background] Tehrani S, Mobarrez F, Antovic A, Santesson P, Lins PE, Adamson U, Henriksson P, Wallen NH, Jorneskog G. Atorvastatin has antithrombotic effects in patients with type 1 diabetes and dyslipidemia. Thromb Res. 2010 Sep;126(3):e225-31. doi: 10.1016/j.thromres.2010.05.023. Epub 2010 Jul 15. PMID 20637495
- [Background] Siljander P, Carpen O, Lassila R. Platelet-derived microparticles associate with fibrin during thrombosis. Blood. 1996 Jun 1;87(11):4651-63. PMID 8639834
- [Derived] Tehrani S, Antovic A, Mobarrez F, Mageed K, Lins PE, Adamson U, Wallen HN, Jorneskog G. High-dose aspirin is required to influence plasma fibrin network structure in patients with type 1 diabetes. Diabetes Care. 2012 Feb;35(2):404-8. doi: 10.2337/dc11-1302. Epub 2011 Dec 6. PMID 22148098